CLINICAL TRIAL: NCT02638805
Title: An Open-Label, Multi-Center, Randomized, Phase 3b Study to Evaluate the Safety and Tolerability of Switching to One of Two Dosing Strategies of ITCA 650 in Patients With Type 2 Diabetes Receiving Stable Doses of Liraglutide
Brief Title: Study of the Safety and Tolerability of Switching to ITCA 650 in Patients With Type 2 Diabetes Receiving Liraglutide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-201
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): ITCA 650 20/60 mcg/day
  Interventions: Drug: ITCA 650 Osmotic Mini Pump 20/60 mcg/day; Drug: Metformin; Drug: Liraglutide
- Group 2 (Experimental): ITCA 650 60 mcg/day
  Interventions: Drug: ITCA 650 Osmotic Mini Pump 60 mcg/day; Drug: Metformin; Drug: Liraglutide

INTERVENTIONS:
Drug: ITCA 650 Osmotic Mini Pump 20/60 mcg/day — ITCA 650 osmotic mini pump delivering exenatide 20/60 mcg/day
  Arms: Group 1
Drug: ITCA 650 Osmotic Mini Pump 60 mcg/day — ITCA 650 osmotic mini pump delivering exenatide 60 mcg/day
  Arms: Group 2
Drug: Metformin — Stable dose for at least 3 months (at least 1000 mg/day)
Drug: Liraglutide — Stable dose for at least 3 months (at least 1.2 mg/day)

SUMMARY:
A Phase 3b, open-label, randomized, multicenter, safety and tolerability study of ITCA 650 in subjects with Type 2 diabetes taking liraglutide and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes ≥ 3 months.
* Stable regimen of diet and exercise in combination with a stable treatment of liraglutide ≥1.2 mg/day and metformin ≥1000 mg/day.
* HbA1c ≤9.5%.
* Stable body weight ≥ 3 months.
* Body mass index (BMI) ≥25 to ≤45 kg per meter squared.
* Calcitonin <50 ng/L (50 pg/mL) at the Screening Visit.

Exclusion Criteria:

* History of type 1 diabetes.
* Recent use or of anti-diabetic medications other than liraglutide or metformin.
* History of significant/severe nausea and/or vomiting due to liraglutide.
* Significant symptomatic hyperglycemia.
* History or evidence, within the last 6 months prior to the Screening Visit, of myocardial infarction, coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention), unstable angina, or cerebrovascular accident or stroke.
* History or evidence of acute or chronic pancreatitis.
* History of liver disease.
* History of medullary thyroid cancer or a family or personal history of multiple endocrine neoplasia type 2.
* Poor thyroid, liver, or renal function.
* Serum creatinine levels >1.5mg/dL (132 μmol/L) for male patients, or >1.4 mg/dL (123 μmol/L) for female patients.
* Weight loss surgery or requires weight loss medications.
* History of malignancy (not including basal or squamous cell carcinoma of the skin with past 5 years).
* History of active alcohol or substance abuse.
* Treatment with medications that affect GI motility.
* History of hypersensitivity to exenatide or liraglutide.
* Women that are pregnant, lactating, or planning to become pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number (percentage) and severity of treatment-emergent adverse events (TEAEs) of nausea and/or vomiting | From Randomization to 34 weeks
  Number (percentage) and severity of treatment-emergent AEs (TEAEs) of nausea and/or vomiting over the 26-week treatment period; treatment discontinuation for nausea and/or vomiting; and pattern of nausea and/or vomiting over time.

SECONDARY OUTCOMES:
Number (percentage) and severity of all treatment-emergent adverse events | From Randomization to 34 weeks
  All TEAEs 2 dose regimens of ITCA 650 over 26 weeks in patients with T2D after switching from stable therapy with liraglutide
Incidence of hypoglycemia | From Randomization to 34 weeks
Change in percentage of glycosylated hemoglobin (HbA1c) in the blood | From baseline to Week 26
Change in body weight | from baseline to Week 26
  Change from baseline in body weight at Week 26

OTHER OUTCOMES:
Change from baseline in blood pressure and heart rate | from baseline to 34 weeks
  Change from baseline in blood pressure and heart rate at Week 26
Change from baseline in fasting plasma glucose | from baseline to Week 26
Change from baseline in cholesterol | from baseline to Week 26
  Change in low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Saint Vincent's Medical Center (BRANY), Gulf Shores, Alabama
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - University of Colorado Hospital, Aurora, Colorado
  - Denver VA Medical Center, Denver, Colorado
  - Meridien Research, Brooksville, Florida
  - International Research Associates, LLC, Hialeah, Florida
  - Care Partners Clinical Research, LLC, Jacksonville, Florida
  - AMPM Research Clinic, Miami, Florida
  - Epocrates Medical and Research Center, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Solaris Clinical Research, Meridian, Idaho
  - American Health Network of Indiana, LLC, Avon, Indiana
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - American Health Network of Indiana, LLC, Greenfield, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Center for Advanced Medical Research, City of Saint Peters, Missouri
  - Radiant Research, St Louis, Missouri
  - Accent Clinical Trials, Las Vegas, Nevada
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Manhattan Medical Research, New York, New York
  - Novel Research of New York, The Bronx, New York
  - Carteret Medical Group, LLC, Morehead City, North Carolina
  - Prestige Clinical Research, Franklin, Ohio
  - Lynn Institute of the Oz, Norman, Oklahoma
  - LION Research, Norman, Oklahoma
  - University of Tennessee Health Sciences Center, Memphis, Tennessee
  - Coastal Bend Clinical Research, Corpus Christi, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Juno Research, LLC, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Panacea Clinical Research, LLC, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Victorium Clinical Research Ltd., San Antonio, Texas
  - Erickson Research and Development, Clinton, Utah

IPD SHARING:
Plan to Share IPD: No